CLINICAL TRIAL: NCT01375439
Title: Maternal and Perinatal Outcome in Women With History of Premature Labor in Previous Pregnancy and Submitted to Active Search of Genital Infection
Brief Title: Maternal and Perinatal Outcome in Women With History of Premature Labor in Previous Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Danielle Cristina Alves Feitosa Gondo, dr, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ddt1333
Record Dates: First submitted 2011-03-23; First posted 2011-06-17 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2011-07

CONDITIONS: Pregnancy; Vulvovaginitis; Uterine Cervicitis; Pregnancy Outcome
Keywords: Pregnancy; vulvovaginitis; uterine cervicitis; pregnancy outcome
MeSH Terms: conditions — Vulvovaginitis; Uterine Cervicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active search of lower genital tract infections (Other): Active search of lower genital tract infections
  Two groups (G1 and G2) will be part of study, each one composed of 140 pregnant women with a history of premature birth, G1 will have the active search and etiologic diagnosis of lower genital tract infections and G2 do not search of these infections, keeping for this group, the protocol of routine care of basic health units in the city of Botucatu. Workup care of pregnant women (G1) will include the completion of direct examination of vaginal contents stained by Gram's method, culture in the medium of Diamonds and polymerase chain reaction (PCR) of endocervical secretions, collected by health services in primary care the municipality in two moments: before 20th pregnancy week (M1) and in 36th pregnancy week (M2). The moment M3 will be after the birth, to evaluate the perinatal outcome.
  Interventions: Other: Active search of lower genital tract infections

INTERVENTIONS:
Other: Active search of lower genital tract infections — Two groups (G1 and G2) will be part of study, each one composed of 140 pregnant women with a history of premature birth, G1 will have the active search and etiologic diagnosis of lower genital tract infections and G2 do not search of these infections, keeping for this group, the protocol of routine care of basic health units in the city of Botucatu. Workup care of pregnant women (G1) will include the completion of direct examination of vaginal contents stained by Gram's method, culture in the medium of Diamonds and polymerase chain reaction (PCR) of endocervical secretions, collected by health services in primary care the municipality in two moments: before 20th pregnancy week (M1) and in 36th pregnancy week (M2). The moment M3 will be after the birth, to evaluate the perinatal outcome.

SUMMARY:
Introduction: Preterm labor (PTL) is an important obstetric intercurrence that affects 5 to 10% of pregnancies. Among the known factors of PTL etiology are PTL occurrence in previous pregnancies, multiple pregnancies, polyhydramnios, vaginal bleeding during pregnancy, premature membrane rupture (PMR) and bacterial vaginosis. Despite the advancement achieved in Neonatology, morbidity and mortality resulting from high rates of preterm births have remained constant in the last few decades. Objective: This study aims at evaluating maternal and perinatal outcomes of pregnant women with a history of preterm labor in previous pregnancies and submitted to active search for vaginal infection. Material and Method: It is a prospective-cohort epidemiological study to be conducted in Botucatu/SP. Two study groups (G1 and G2) will be formed, and each of them will comprise 140 pregnant women with a history of preterm childbirth. G1 will be related to the active search and etiological diagnosis of lower genital tract infections, and G2 will be related to non-search for such infections, for which the routine care protocol of primary health units in the city of Botucatu will be maintained. Care propedeutics for the pregnant women (G1) will include the performance of direct examination of vaginal content stained by the Gram method, culture in Diamonds medium, polymerase chain reaction (PCR) of endocervical secretion collected in the primary health care services in the city at two moments: prior to the 20th gestational week (M1) and at the 36th week (M2). Moment M3 will take place after childbirth for evaluation of the perinatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in the study women with a history of preterm labor in previous pregnancy, without other risk factors identified in the initial prenatal current to initiate prenatal care until 20 weeks of gestation in any unit of primary care and Botucatu they have agreed to participate.

Exclusion Criteria:

* Will be excluded from the study women who have complications during pregnancy such as urinary tract infections, severe periodontal disease, hypertension, diabetes or multiple gestation, among others.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Track pregnant women priority for the exams that allow the etiologic diagnosis of lower genital tract infections. | Up to 6 months after birth
  This study starts from the assumption that the active search and etiologic treatment of genital infections can reduce adverse pregnancy outcome and, if confirmed, could subsidize health managers in the implementation of actions aimed at introducing, in the health services of varying degrees of complexity , the etiologic diagnosis of lower genital tract infections. It is known that the costs of such a diagnosis are high and could have prevented the routine examination of patients during prenatal care.